CLINICAL TRIAL: NCT00384124
Title: Phase III Trial of 6 Weeks of Imiquimod for the Treatment of Bowens Disease of the Head and Neck. Outcome is Histologic Clearance at 14 Weeks.
Brief Title: Topical Imiquimod for Bowen's Disease of the Head and Neck
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Nicole Owens, MD, Brooke Army Medical Center Department of Dermatology
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C.2005.087
Record Dates: First submitted 2006-10-04; First posted 2006-10-05 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Bowens Disease
Keywords: Bowens disease; Squamous cell carcinoma in situ of the skin; imiquimod
MeSH Terms: conditions — Bowen's Disease | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Imiquimod — Imiquimod application M-F for six weeks (total of 30 applications) followed by surgical excision of site
  Other Names: Aldara

SUMMARY:
* Double blinded, randomized, placebo controlled trial of imiquimod for the treatment of histologically proven Bowens disease of the head and neck.
* Null hypothesis: No difference in histologic clearance rates of patients with head or neck Bowens treated with imiquimod versus placebo.
* Outcome: Histologic clearance of Bowens disease at T=14 weeks.

DETAILED DESCRIPTION:
Interventional study Enrolling

Inclusion criteria: Military beneficiaries with histologically proven Bowens disease, located on the head and neck, defined as any area superior to the clavicle and anterior to the posterior triangle of the neck

Exclusion Criteria:

* Previous treatment of biopsied lesion Recurrent lesions from previous biopsy-proven Bowen's disease
* Patients younger than 18 years of age
* Pregnancy
* Immunosuppression, including HIV, transplant patients on immune suppressive medications, cancer patients on chemotherapy, and hematologic malignancies (e.g., lymphoma, leukemia)
* Mucous membrane involvement
* Lesions larger than 2 cm

  * Methods: Pts randomized to treatment group (6 weeks of Mon-Friday Imiquimod to Bowens site) or vehicle group (same treatment regimen). All patients undergo surgical excision (Mohs or simple excision) of site where disease is either visible or was present and tissue examined for histologic evidence of residual Bowens disease

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of Bowen's disease (squamous cell carcinoma in situ), defined as full-thickness keratinocyte atypia and architectural disorder limited to the epidermis, with or without involvement of the follicular unit

  * Located on the head and neck, defined as any area superior to the clavicle and anterior to the posterior triangle of the neck
  * Primary Bowen's disease (first diagnosis)

Exclusion Criteria:

* Previous treatment of biopsied lesion
* Recurrent lesions from previous biopsy-proven Bowen's disease
* Patients younger than 18 years of age
* Pregnancy
* Immunosuppression, including HIV, transplant patients on immune suppressive medications, cancer patients on chemotherapy, and hematologic malignancies (e.g., lymphoma, leukemia)
* Mucous membrane involvement
* Lesions larger than 2 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
histologic clearance of Bowens disease in treated versus placebo group | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicole M Owens, MD, Principal Investigator — Brooke Army Medical Center Department of Dermatology
Locations (1):
- Brooke Army Medical Center Department of Dermatology, Fort Sam Houston, Texas, United States